CLINICAL TRIAL: NCT03695913
Title: Continuous Glucose Monitoring With a Low Carbohydrate Diet to Reduce Weight in Patients With Pre-Diabetes
Brief Title: Continuous Glucose Monitoring (CGM) With a Low Carbohydrate Diet to Reduce Weight in Patients With Pre-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Caroline Richardson, Dr Max and Buena Lichter Research Professor of Family Medicine, Assistant Chair, Department of Family Medicine and Professor of Family Medicine, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00145667
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Pre-diabetes
Keywords: Pre-diabetes, low carbohydrate diet
MeSH Terms: conditions — Glucose Intolerance | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Normal Diet + CGM then low carb + CGM (Experimental): Phase I (part 1) - regular diet:
  Patients will wear a CGM sensor (with no real time feedback) for 11 days; document what they eat on a food log; and rate their postprandial fatigue and cravings.
  Phase II (part 2) - low carb diet:
  Patients will wear a CGM sensor (with real time feedback) for 11 days; document what they eat on a food log; and rate their postprandial fatigue and cravings; document their blood sugar before and two hours after eating (as well as before breakfast and before going to bed).
  Interventions: Other: Normal Diet; Other: Low carb diet; Device: CGM with no real time feedback; Device: CGM with real time feedback); Behavioral: Education material

INTERVENTIONS:
Other: Normal Diet — Phase I (regular diet):
  all participants will eat their normal diet and will log their food.
Other: Low carb diet — Phase II (low carb diet):
  participants will be asked to eat a low carb diet and log their food
Device: CGM with no real time feedback — Phase I will collect CGM without real time feedback
Device: CGM with real time feedback) — Phase II participants will be asked to scan their sensor at least every eight hours and document their blood sugar before and two hours after eating as well as before breakfast and before going to bed.
Behavioral: Education material — Phase I: participants will be given the book Always Hungry and be asked to read chapters 1-5 after a health check phone call approximately 5 days after the sensor is placed.
  Phase II: participants will be taught about carbohydrates and the benefits and side effects. Additionally, they will be given multiple resources to assist them regarding carbohydrates as well as a book entitled "The Calorie King, Calories, Fat, and Carbohydrates." Groceries will also be delivered for 2 recipes that the participants choose from to make.

SUMMARY:
This study will recruit pre-diabetic patients to see if continuous glucose monitoring (CGM) with a low carbohydrate diet can reduce the percentage of time the CGM readings are above the normal range. Through this study it will demonstrate the feasibility of using CGM with a low carbohydrate diet to reduce weight and risk of developing diabetes in patients with pre-diabetes.

Patients that appear to be eligible will be recruited from Michigan Medicine in the Family Medicine Clinic at the Livonia Center.

ELIGIBILITY:
Inclusion Criteria:

* A1C Glucose Measurement between 5.7 to 6.4 (for most recent A1C test, not older than 1 year)
* No diabetes medication including Metformin
* BMI (body mass index) >30
* Must speak, read, and write in English
* No current pregnancy or breastfeeding
* Must not classify as either Vegan or Vegetarian
* Must be a patient at the Livonia Health Center

Exclusion Criteria:

* previous bariatric surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Richardson, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Livonia, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Diet + CGM, Then Low Carb + CGM: For 11 days, patients will wear a CGM sensor (with no real time feedback), eat a regular diet, document what they eat on a food log and rate their postprandial fatigue and cravings. Then, for 11 days, patients will eat a low-carb diet, wear a CGM sensor (with real time feedback), document what they eat on a food log, rate their postprandial fatigue and cravings, and document their blood sugar before and two hours after eating (as well as before breakfast and before going to bed).
Period: Overall Study
Arm/Group | Normal Diet + CGM, Then Low Carb + CGM
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Diet + CGM Then Low Carb + CGM: For 11 days, patients will wear a CGM sensor (with no real time feedback), eat a regular diet, document what they eat on a food log and rate their postprandial fatigue and cravings. Then, for 11 days, patients will eat a low-carb diet, wear a CGM sensor (with real time feedback), document what they eat on a food log, rate their postprandial fatigue and cravings, and document their blood sugar before and two hours after eating (as well as before breakfast and before going to bed).
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Knowledge of Low Carbohydrate Eating [Mean (Standard Deviation); unit: score on a scale] — The Low Carbohydrate Knowledge Scale ranges from 1 to 30, where 1 is a low score and 30 is a high score. Population: One participant did not complete the baseline survey
  score on a scale
    number analyzed (Participants) | 14
    (all) | 26.4 (1.65)

OUTCOME MEASURES:

1. Primary Outcome: Participant Satisfaction With Continuous Glucose Monitoring (CGM)
Description: Satisfaction is measured using responses to the post intervention survey question, "How likely are you to recommend that a friend or family member with pre-diabetes wear a continuous glucose monitor (CGM)?". A 5 point scale was used, ranging from 1 to 5, where a score of 1 is "extremely likely" and 5 is "would not recommend". Satisfied respondents answered either 1 or 2 on the scale.
Time Frame: 33 days after day 1 (visit 3 completion)
Measure: Number; unit: participants
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
participants
  1 - extremely likely | 10
  2 - likely | 4
  3- Neither likely or unlikely | 1
  4 - Not likely | 0
  5 - Would not recommend | 0

2. Primary Outcome: Participant Satisfaction With Continuous Glucose Monitoring
Description: Common qualitative themes related to participant satisfaction with CGM from post intervention interview were coded.
Time Frame: 60 days (30 days after visit 3 completion)
Population: 2 participants did not participate in the qualitative interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 13
Participants
  Respondents perceived no barriers to CGM use | 13
  Respondents attempted the low carb diet | 13

3. Secondary Outcome: Feasibility, Measured by Recruitment
Description: Successful recruitment completed within 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
Participants | 15

4. Secondary Outcome: Feasibility of Pre-diabetic Patients to Wear CGM Sensors
Description: Feasibility is measured by the number of participants who wore a sensor for at least 20 out of 22 days
Time Frame: completed within 60 days of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
Participants | 15

5. Secondary Outcome: Weight Change
Description: Change between visit 1 and the final visit.
Time Frame: day 11 (visit 2), day 22 (visit 3)
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
pounds | -1.41 (2.18)

6. Secondary Outcome: Change in Percentage of Time Glucose is Above 140
Description: Comparison between the first sensor wear period and the second sensor wear period.
Time Frame: 33 days after day 1
Measure: Mean (Standard Deviation); unit: Percentage of Time Glucose is 140+
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 14
Percentage of Time Glucose is 140+ | -2.6 (6.5)

7. Secondary Outcome: Number of Participants Who Reported Side Effects of Low Carbohydrate Eating and CGM at Health Check Phone Call
Description: During the health check phone call survey, participants were asked to report whether they experienced any side effects.
Time Frame: Approximately 5 days each new sensor is placed (days 5 and 16)
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
Participants | 0

8. Secondary Outcome: Number of Participants Who Reported Side Effects of Low Carbohydrate Eating and CGM in Patient Log
Description: In the patient side effect log, participants recorded whether they experienced any side effects.
Time Frame: days 11 through 22
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
Participants | 1

9. Secondary Outcome: Change in Knowledge of Low Carbohydrate Eating
Description: The Low Carbohydrate Knowledge Scale ranges from 15-41, where 15 is a low score and 41 is a high score. Participants were asked to report knowledge at baseline and completion. A positive score indicates an increase from baseline in knowledge, while a score of 15 indicates no change and a negative score indicates a decrease in knowledge from baseline.
Time Frame: baseline, day 22
Population: One participant did not complete the baseline survey, so change could not be assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 14
score on a scale | .57 (1.34)

10. Secondary Outcome: Change in Cravings From Day 11 to Day 22
Description: Participants recorded cravings in food logs. Craving rating scale ranges from 1 to 5, where a score of 1 is low and a score of 5 is high.
Time Frame: 11 days
Population: 10 participants submitted both pre- and post-intervention food logs. Data was unusable for 5 participants because they either did not complete the pre-intervention food log and/or they didn't complete the post-intervention food log
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 10
score on a scale | -.625 (.93)

11. Secondary Outcome: Intention to Continue Low Carbohydrate Eating
Description: The completion survey asked participants a question, "How confident are you that you can maintain a low carbohydrate diet for the next 12 months?" Intention to Continue Low Carbohydrate eating used a scale of 1 to 5, where a score of 1 was not confident at all and a score of 5 was very confident.
Time Frame: day 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
score on a scale | 4.5 (.51)

12. Secondary Outcome: Utility of CGM Feedback for Changing Diet
Description: Utility of CGM feedback is expressed as the number of participants who qualitatively indicated that CGM feedback helped them to change their diet. Themes were identified and coded from qualitative interviews around this topic. Two qualitative coders identified themes that supported this construct.
Time Frame: 60 days (30 days after visit 3 completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Normal Diet + CGM Then Low Carb + CGM
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Diet + CGM Then Low Carb + CGM (N=15)
Bleeding at Insertion site (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This was a small pilot study to test feasibility of CGM. No statistical analysis was conducted because of the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT03695913/Prot_000.pdf